CLINICAL TRIAL: NCT03137927
Title: A Phase I Clinical Study of a GamLPV, a Live Intranasal Bordetella Pertussis Vaccine; A Randomized Placebo-controlled Dose-escalating Study of Single-use GamLPV Safety and Tolerability in Healthy Human Volunteers
Brief Title: A Phase I Clinical Study of a GamLPV, a Live Intranasal Bordetella Pertussis Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GamLPV-01
Record Dates: First submitted 2017-04-25; First posted 2017-05-03 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-04

CONDITIONS: Whooping Cough
Keywords: bordetella pertussis; vaccine; Immunologic Factors; whooping cough
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Intervention Model Description: The study is dose-escalating, so there will be 3 groups. Group 1: 9 individuals will be vaccinated intranasally with 2,5*108 bacteria (CFU), 3 individuals will get placebo.
  Group 2: 9 individuals will be vaccinated intranasally with 109 bacteria cells(CFU), 3 individuals will get placebo.
  Group 3: 9 individuals will be vaccinated intranasally with 4*109 bacteria cells(CFU), 3 individuals will get placebo.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 Vaccine GamLPV (Experimental): 9 individuals will be vaccinated intranasally with 2,5*10*8 bacteria cells (CFU)
  Interventions: Biological: Vaccine GamLPV
- Group 1 placebo (Placebo Comparator): 3 individuals will get placebo
  Interventions: Other: Placebo
- Group 2 Vaccine GamLPV (Experimental): 9 individuals will be vaccinated intranasally with 10*9 bacteria cells(CFU)
  Interventions: Biological: Vaccine GamLPV
- Group 2 placebo (Placebo Comparator): 3 individuals will get placebo
  Interventions: Other: Placebo
- Group 3 Vaccine GamLPV (Experimental): 9 individuals will be vaccinated intranasally with 4*10*9 bacteria cells(CFU)
  Interventions: Biological: Vaccine GamLPV
- Group 3 placebo (Placebo Comparator): 3 individuals will get placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Vaccine GamLPV — live intranasal vaccine for whooping cough prevention
  Other Names: live intranasal Bordetella pertussis vaccine
  Arms: Group 1 Vaccine GamLPV; Group 2 Vaccine GamLPV; Group 3 Vaccine GamLPV
Other: Placebo — Placebo
  Arms: Group 1 placebo; Group 2 placebo; Group 3 placebo

SUMMARY:
The study contains three periods: screening, inpatient hospitalization and follow-up. And should be leaded as a randomized placebo-controlled study with in chain order enrolled volunteers and dose escalating.

DETAILED DESCRIPTION:
After screening, verifying of inclusion/exclusion criteria and signing of informed consent statement volunteers will be directed in a hospital and hospitalized in individual boxes.

Vaccine (GamLPV) or placebo will be administered to groups of volunteers. Each group includes 12 individuals. The study is dose-escalating, so there will be 3 groups.

Group 1: 9 individuals will be vaccinated intranasally with 2,5*108 bacteria (CFU), 3 individuals will get placebo.

Group 2: 9 individuals will be vaccinated intranasally with 109 bacteria cells(CFU), 3 individuals will get placebo.

Group 3: 9 individuals will be vaccinated intranasally with 4*109 bacteria cells(CFU), 3 individuals will get placebo.

On the third day volunteers will be discharged from hospital. 4 visits will be held during outpatient observation- on 8, 15, 29 and 60 days after administration - for physical examination and laboratory assessment. Beside that it would be suggested to volunteers to extend a deadline of participation in the clinical study until 150-th day.

For each dosing group the consecutive inclusion of volunteers with the intermediate evaluation of the safety parameters is stipulated. The group (12 people) is divided into two parts. Originally the first part (5 volunteers) is included in the study. Randomization will be performed by choosing the envelope with the randomizing number at the day of hospitalization. The volunteer will be given either the investigating laboratory specimen or placebo. The researcher includes in the study the 2nd part of the group (7 people) after the evaluation of the intermediate results of the safety analyses (total blood count, biochemical analysis, urinalysis, general examination of a patient). The researcher compiles the intermediate report with the analysis of the endurance of the investigating dose of the preparation after the evaluation of the intermediate safety results. The criterion of the endurance and the dose safety will be at first the absence of serious undesirable phenomena and clinically important shifts of the laboratory indices connected with the administration of the investigating preparation. The decision about the advisability to continue the study and to pass to the 2nd part of volunteers and (or) to escalate the dose will be made by the "Independent committee for data monitoring (ICDM) for periodical examination of the clinical study, safety data and/or main parameters of the efficacy" as well it must be approved by the Local/Independent Ethical Committee of the Research centerе.

After getting the permission to continue the study the next group will be organized according to the analogous scheme: at first the first group of volunteers and then, after receiving the safety results in a written form, the 2nd group will be included, the decision to pass from the second group to the third will be the same.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females within the age range from 18 to 40 years
2. Health physical condition must be confirmed by routine clinical, laboratory and instrumental methods of diagnosis (absence of gastrointestinal, renal, cardiovascular diseases, hepatic, blood disorders, cancer and infectious diseases)
3. Body-weight index within range from 18 to 30 kg\m2
4. Consent for using of reliable contraception (contraception sheath with spermicidal agents) while study and three months after the end of the study
5. Signed Participant Information Sheet and informed consent
6. Absence of specific antibodies (IgG, IgM, IgA) to Bordetella pertussis (negative ELISA results according to direction for ELISA test-system)
7. Absence of Bordetella pertussis DNA in nasopharyngeal swabs (negative PCR results)

Exclusion Criteria:

1. Whooping cough in past medical history
2. Vaccination against whooping cough over the past decade
3. Any other anti-infective immunization during last year
4. Any medical condition (renal diseases, hepatic disorders, haematological malignancies, malignant neoplasms and other diseases) which, in the opinion of the investigator, might interfere with the evaluation of the study objectives
5. Vaccine-associated diseases or clinically significant vaccinal reactions in medical history
6. Clinically significant abnormal laboratory values at the discretion of the investigator
7. Use of any medications (in particular herbal medications and dietary supplements) within 30 days after day 0 at the discretion of the investigator
8. Positive results of HIV, hepatitis B or C
9. Use of narcotic drugs and/or a history of drug/alcohol abuse
10. Allergic diseases in medical history (in particular drug reaction and food allergy)
11. The subject has donated blood/plasma or suffered from blood loss of at least 450 ml (1 unit of blood) within 6 weeks prior to screening
12. Current participation in any other clinical trial or participation (and during the whole study) in any clinical trial in the previous 3 months prior to day 0
13. Inability to adhere to the protocol
14. Acute infectious diseases within 4 weeks prior to screening
15. Wheezing on the results of peakflowmetry
16. Significant ECG changes
17. Pregnancy or lactation (for female volunteers)
18. Systolic blood pressure less than 90 mmHg or over than 130 mmHg; diastolic blood pressure less than 60 mmHg or over 90 mmHg
19. Heart rate less than 60 bpm or more than 90 bpm

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | the total Time Frame is 150 days after the vaccination
  Evaluation of general safety and tolerability of medicinal product "GamLPV, a live intranasal vaccine for whooping cough prevention" in healthy human volunteers compared to placebo, detection the most frequent from possible adverse events of GamLPV

SECONDARY OUTCOMES:
Dose ranging and optimal dose choice | the total Time Frame is 150 days after the vaccination
  Dose ranging and optimal dose choice for safety and tolerability of medicinal product GamLPV, a live intranasal vaccine for whooping cough prevention" in further clinical trials
specific antibody response to B.pertussis | the total Time Frame is 150 days after the vaccination
  • To assess specific antibody response to B.pertussis after vaccination by "GamLPV, a live intranasal vaccine for whooping cough prevention"
dynamics of bacteria generation in nasopharynx of human volunteers | the total Time Frame is 150 days after the vaccination
  To see if the attenuated B.pertussis bacteria have the ability to colonise the human respiratory tract after vaccination by "GamLPV, a live intranasal vaccine for whooping cough prevention" and to assess dynamics of bacteria generation in nasopharynx of human volunteers
the B- and T-cell immune responses to B.pertussis | the total Time Frame is 150 days after the vaccination
  To assess the B- and T-cell immune responses to B.pertussis in response to vaccination by "GamLPV, a live intranasal vaccine for whooping cough prevention"

CONTACTS AND LOCATIONS:
Overall Officials: Marina Rusanova, Principal Investigator — Infectious Disease Clinical Hospital No. 1 of the Moscow Healthcare Department
Locations (1):
- Infectious Disease Clinical Hospital No. 1 of the Moscow Healthcare Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided